CLINICAL TRIAL: NCT04614259
Title: Perioperative Pain Management for Cleft Lip Repair in Children, Bilateral Infraorbital Nerve Block Versus Conventional Methods( Combined IV Fentanyl With Peri Incisional Infiltration). A Randomized Comparative Study
Brief Title: Perioperative Pain Management for Cleft Lip in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Elsonbaty, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N 49-2018/Ms
Record Dates: First submitted 2020-10-21; First posted 2020-11-03 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Perioperative Complication Pain
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intravenous analgesia (Experimental)
  Interventions: Combination Product: i.v. analgesia
- infraorbital nerve block (Experimental)
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — The infraorbital foramen was located at the floor of the orbital rim at about the level of the pupil,The upper lip was folded back and a finger is placed externally at the level of the infraorbital foramen to prevent the needle from the cephalad insertion in the globe of the eye. A 27-gauge needle was bent about 70 degree to ease the insertion through the buccal mucosa over the maxillary process, towards the infraorbital foramen.
  After careful aspiration the local anesthetic was injected (injection of 3 ml 0.25% bupivacaine in 1:200.000 adrenaline ,1.5 ml on each side). [104] Pressure was needed to be applied for one minute to the area as there is loose adventitious tissue that can lead to swelling and ecchymosis
  Arms: infraorbital nerve block
Combination Product: i.v. analgesia — Using inhalational induction with sevoflurane as tolerated , atracurium 0.5mg/kg to facilitate endotracheal intubation and fentanyl 1 mcg/kg ,Mechanical ventilation was adjusted to maintain 30 to 35 mmHg end-tidal carbon dioxide, anesthesia was maintained with 1.5 % isoflurane and atracurium (0.1 mg/kg every 30 minutes) ,all patients were received intraoperative diclofenac sodium 0.5 mg/kg intramuscular .
  Blood pressure and heart rate were measured 5 minutes after endotracheal intubation and every 15 minutes till recovery from the anesthesia then every 15 min in the postoperative care unite for 30 minutes
  Arms: intravenous analgesia

SUMMARY:
Single blind prospective randomized comparative study. 76 children between 6 months and 3 years with cleft lip will be divided in two groups. 38 children group C conventional group and 38 children group S infraorbital nerve block group.

ELIGIBILITY:
Inclusion Criteria:

* good physical condition.
* Age 6 months to 3 years.
* Scheduled to undergo operations for cleft lip repair. Genders eligible for study are both .

Exclusion Criteria:

* Children posted for combined procedures like congenital heart correction with palatoplasty .
* Parents refusal .
* Bleeding disorders( platelets count < 100.000 , international ratio >1.5).
* Skin lesions or wounds at site of needle insertion .
* Co-morbidities as congenital heart disease , lung pathology or central nervous system
* Known hypersensitivity to local anesthetics or opioids .

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 24 huors
  Total rescue doses of morphine

IPD SHARING:
Plan to Share IPD: No
Do not share

REFERENCES:
- [Background] Pain terms: a list with definitions and notes on usage. Recommended by the IASP Subcommittee on Taxonomy. Pain. 1979 Jun;6(3):249. No abstract available. PMID 460932
- [Background] Lee SJ, Ralston HJ, Drey EA, Partridge JC, Rosen MA. Fetal pain: a systematic multidisciplinary review of the evidence. JAMA. 2005 Aug 24;294(8):947-54. doi: 10.1001/jama.294.8.947. PMID 16118385
- [Background] Tremlett M. Anaesthesia for cleft lip and palate surgery. Curr Anaesth Crit Care. 2004;15:309-16.
- [Background] Doyle E, Hudson I. Anesthesia for primary repair of cleft lip and cleft palate: a review of 244 procedures. Paediatr Anaesth 1992; 2: 139-145.
- [Background] Takemura H, Yasumoto K, Toi T, Hosoyamada A. Correlation of cleft type with incidence of perioperative respiratory complications in infants with cleft lip and palate. Paediatr Anaesth. 2002 Sep;12(7):585-8. doi: 10.1046/j.1460-9592.2002.00906.x. PMID 12358652